CLINICAL TRIAL: NCT06398691
Title: Is it Possible to Premature Newborns Treated With Less Invasive Surfactant Administration Under Heated Humidified High-flow Air With Nasal Cannula?
Brief Title: Premature Newborns Treated With Less Invasive Surfactant Administration Under Heated Humidified High-flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, MELEK BUYUKEREN, Associate Professor, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU-MB-1
Record Dates: First submitted 2024-03-15; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Disease; Newborn Rds
Keywords: NEWBORN; Respiratory Distress Syndrome; Less Invasive Surfactant Administration; Heated Humidified High-Flow Air Support with Nasal Cannula.; Nasal Continuous Airway Pressure
MeSH Terms: conditions — Respiration Disorders; Pulmonary Atelectasis; Respiratory Distress Syndrome | interventions — Cannula

STUDY DESIGN:
Intervention Model Description: Premature newborns (gestational age <370/7 weeks) who did not require intubation, who were diagnosed with RDS, and who were treated with surfactant in the first 72 hours of life were included in the study. Written informed consent was obtained from all of the infants' families before the infants were enrolled in the study. Noninvasive respiratory support was provided by nasal CPAP or HHHNFC, respectively, according to the time of admission to the intensive-care unit, so the patients were divided into two groups. During the study period, the noninvasive respiratory support method (nasal CPAP or HHHNFC) that the babies received did not change.
  Post-hoc, one-way difference between two independent means (two groups) statistical analysis was used. Significance P < 0.05; effect size 0.9; power (1-ß err prob) was found to be 82%.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP group (Active Comparator): A Babylog 8000 neonatal ventilator (Dräger, Lübeck, Germany) for nasal CPAP support was used support . The nasal CPAP support had been applied through short binasal prongs (Optiflow Junior 2 nasal cannula) used as an interface. PEEP pressure was set to 6-8 cmH2O for nasal CPAP. The FiO2 was regulated to keep the oxygen-saturation value between 92% and 95%.
  Interventions: Device: Nazal CPAP
- HHHFNC group (Active Comparator): A Vapotherm® device (Vapotherm Inc., Stevensville, MD) for HHHFNC support was used. The airflow rate was set to 6-8 L/min for HHHFNC (heat: 37 °C). The HHHFNC support had been applied through the small bore cannula in the Vapotherm as an interface. The FiO2 was regulated to keep the oxygen-saturation value between 92% and 95%.
  Interventions: Device: Heated humidified high-flow air support with nasal cannula

INTERVENTIONS:
Device: Nazal CPAP
  Arms: CPAP group
Device: Heated humidified high-flow air support with nasal cannula
  Arms: HHHFNC group

SUMMARY:
Nasal Continuous Airway Pressure (CPAP) or Heated humidified high-flow Air support with nasal cannula (HHHFNC) are among the most commonly used non-invasive respiratory support methods. The purpose of this prospective study was to compare vital findings, blood gas parameters, perfusion index (PI) and plethysmographic variability index (PVI) values in premature infants treated with less invasive surfactant administration (LISA) under HHHFNC or CPAP.

DETAILED DESCRIPTION:
Nasal Continuous Airway Pressure (CPAP) or Heated humidified high-flow Air support with nasal cannula (HHHFNC) are among the most commonly used non-invasive respiratory support methods. The purpose of this prospective study was to compare vital findings, blood gas parameters, perfusion index (PI) and plethysmographic variability index (PVI) values in premature infants treated with less invasive surfactant administration (LISA) under HHHFNC or CPAP. This study was carried out in Hacettepe University Hospital NICU between January and December 2017. Premature newborns who were on noninvazive respiratory support and were diagnosed as RDS within first 72 hours of life, were taken into the study. Noninvasive respiratory support was provided with nasal CPAP or HHHNFC. Pulse oxymetry measurements were obtained before and 5th, 30th, 60th, 120th , 360th minutes, blood gas analysis was performed immediately before and 120th, 360th minutes after surfactant administration.

Post-hoc, one-way difference between two independent means (two groups) statistical analysis was used. Significance P < 0.05; effect size 0.9; power (1-ß err prob) was found to be 82%.

ELIGIBILITY:
Inclusion Criteria:

* Does not require intubation,
* Diagnosed with RDS
* Premature newborns receiving surfactant therapy in the first 72 hours of life
* Those whose families give written consent

Exclusion Criteria:

* Babies whose families do not give written consent
* Newborns diagnosed with early neonatal sepsis
* Newborns with inotropic requirements
* Neonates with hemodynamically significant PDA
* Babies of diabetic mothers
* Babies with a major congenital anomaly
* Newborns with hemodynamic instability,
* Those requiring endotracheal intubation,
* NEC (Stage 2 or higher),
* Those showing ICH (Stage 2 or higher)
* Babies with perfusion disorders in the first three days

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Investigation of the effect of surfactant treatment on the p02 value in blood gases using the LISA method in premature babies with spontaneous breathing during different respiratory support. | 360 minutes after surfactant treatment
  A total of 34 premature babies were included in the study. There were 22 patients in the CPAP group and 12 patients in the HHHFNC group. It was planned to make a comparison between CPAP and HHHNFC groups in terms of bloog gas parameters before, during and after surfactant treatment. Blood gas analysis was performed immediately before and 120th, 360th minutes after surfactant administration. p02 values in blood gas were determined according to the routine protocol of our NICU. They were performed three times: immediately before the surfactant treatment and at the 120th and 360th minute after the surfactant was administered.

SECONDARY OUTCOMES:
Investigation of the effect of using surfactant treatment with the LISA method during different respiratory support on the pulse oximetry parameters of babies. | 360 minutes after surfactant treatment
  Pulse oxymetry measurements (perfusion index and plethysmographic variability index) were obtained before and 5th, 30th, 60th, 120th , 360th minutes.Masimo Radical-7® Pulse CO-Oximetry (Masimo Corp., Irvine, CA, USA) devices were used. Pulse oximeters were attached to the right wrist of all patients during the study, and preductal measurements were made. The PI and PVI records were taken when the plethysmograph pulse wave was artefact free, while the baby was calm. All vital findings were noted simultaneously. The measurements recorded for six hours after the surfactant administration were transferred to a personal computer and analyzed with the VitaWin 3 (Telematya Germany, Teltow, Germany) program.

CONTACTS AND LOCATIONS:
Overall Officials: MELEK BUYUKEREN, Study Director — Hacettepe University, Neonatology
Locations (1):
- Melek Büyükeren, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, clinical study report
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Result] Morley CJ, Davis PG, Doyle LW, Brion LP, Hascoet JM, Carlin JB; COIN Trial Investigators. Nasal CPAP or intubation at birth for very preterm infants. N Engl J Med. 2008 Feb 14;358(7):700-8. doi: 10.1056/NEJMoa072788. PMID 18272893
- [Result] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GH, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2016 Update. Neonatology. 2017;111(2):107-125. doi: 10.1159/000448985. Epub 2016 Sep 21. PMID 27649091
- [Result] Chao KY, Chen YL, Tsai LY, Chien YH, Mu SC. The Role of Heated Humidified High-flow Nasal Cannula as Noninvasive Respiratory Support in Neonates. Pediatr Neonatol. 2017 Aug;58(4):295-302. doi: 10.1016/j.pedneo.2016.08.007. Epub 2017 Jan 17. PMID 28223010